CLINICAL TRIAL: NCT04557748
Title: Symptoms of Lower Urinary Tract Dysfunction Research Network (LURN) Urinary Urgency Phenotyping Protocol
Brief Title: LURN: Urinary Urgency Phenotyping Protocol
Status: Active, not recruiting | Type: Observational
Sponsor: Arbor Research Collaborative for Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Michigan (Other); Northwestern University (Other); Duke University (Other); University of Iowa (Other); University of Washington (Other); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: LURN 2; U01DK099879 (NIH); U01DK097780 (NIH); U01DK097772 (NIH); U01DK097779 (NIH); U01DK099932 (NIH); U01DK100011 (NIH); U01DK100017 (NIH)
Record Dates: First submitted 2020-09-08; First posted 2020-09-22 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: Lower Urinary Tract Symptoms; Bladder Symptoms; Overactive Bladder; Urinary Urgency; Lower Urinary Tract Dysfunction
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Urinary Bladder, Overactive | interventions — Watchful Waiting; Central Nervous System Sensitization; Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood Serum Plasma Urine Dried blood spots
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- Prospective Observational Cohort Study: Men and women with lower urinary tract symptoms.
  Interventions: Other: Observational
- Prospective Observational Cohort Study Controls: Men and women who do not have urinary dysfunction.
  Interventions: Other: Observational Controls
- Central Sensitization Study: Men and women enrolled in the Prospective Observational Cohort Study with urinary urgency.
  Interventions: Other: Central Sensitization
- Central Sensitization Study Controls: Men and women enrolled in the Prospective Observational Cohort Study with no symptoms of urinary urgency.
  Interventions: Other: Central Sensitization
- Physical Activity and Sleep Study: Men and women enrolled in the Prospective Observational Cohort Study with urinary urgency.
  Interventions: Other: Physical Activity and Sleep Tracker
- Physical Activity and Sleep Study Controls: Men and women enrolled in the Prospective Observational Cohort Study with no symptoms of urinary urgency.
  Interventions: Other: Physical Activity and Sleep Tracker Controls
- Organ-Based Study: Women enrolled in the Prospective Observational Cohort Study with urinary urgency, with and without urgency incontinence.
  Interventions: Other: Organ-Based
- Organ-Based Study Controls: Women enrolled in the Prospective Observational Cohort Study with no symptoms of urinary urgency pr urgency incontinence.
  Interventions: Other: Organ-Based
- Qualitative Assessment of Patients with Urinary Urgency Study: Men and women enrolled in the Prospective Observational Cohort Study with urinary urgency who have treatment plans prescribed at the baseline visit.
  Interventions: Other: Qualitative Assessment of Patients with Urinary Urgency

INTERVENTIONS:
Other: Observational — Treatment:
  Up to five interactions: In-person visits at Baseline, 3 months, and 12 months after initial visit, and phone/online interaction at 6 months and 9 months after initial visit.
  Each in-person follow up visit is expected to last up to 2 hours and each phone/online interaction is expected to last up to 1½ hours.
  Answering questions about your general health and urinary symptoms - may be done remotely Physical exam Completing Self- Reported Measures questionnaires - may be done remotely Completing voiding/intake and food diaries, either online or on paper Weekly text message survey regarding symptom and treatment changes
  Biosample collection:
  At baseline: Up to 4 tablespoons of whole blood, dried blood spots, and urine At baseline: Whole blood will be collected with other biospecimens At 3 months: Up to 4 tablespoons of blood, dried blood spots and urine At 12 months: Dried blood spots
  Groups: Prospective Observational Cohort Study
Other: Observational Controls — One in-person visit that is expected to last up to 2 hours Answering questions about your general health and urinary history Physical exam Completing Self- Reported Measures questionnaires Completing voiding/intake and food diaries, either online or on paper Biosample collection of up to 4 tablespoons of whole blood, dried blood spots, and urine
  Groups: Prospective Observational Cohort Study Controls
Other: Central Sensitization — One in-person visit expected to take up to 30 minutes, that include:
  Segmental Mechanical Hyperalgesia - a hand-held device with a small flat rubber surface will be placed above the pubic bone and forearm, and will apply pressure. Participant will be asked about the intensity and unpleasantness that they experience.
  Pinprick Temporal Summation - participant will receive tactile stimulation by a pointed skin probe ("pinprick stimulator") being placed above the pubic bone and forearm. Participant will be asked to rate the sensation they are feeling.
  Current treatment information including prior surgery or procedures, medication use, other current treatment/therapy used at the time of the visit.
  Self-reported measures questionnaires
  Groups: Central Sensitization Study; Central Sensitization Study Controls
Other: Physical Activity and Sleep Tracker — A physical activity and sleep monitor (Fitbit Charge 3 or similar) will be worn for a 2 week period starting at baseline prior to treatment and again at 3 months. During each 2 week period:
  The Fitbit will be worn both day and night to collect the most information. Text message reminders to wear the Fitbit will be sent. Daily text messages asking the number of nighttime voids you had.
  Groups: Physical Activity and Sleep Study
Other: Physical Activity and Sleep Tracker Controls — A physical activity and sleep monitor (Fitbit Charge 3 or similar) will be worn for a 2 week period at baseline prior to treatment. During the 2 week period:
  The Fitbit will be worn both day and night to collect the most information. Text message reminders to wear the Fitbit will be sent. Daily text messages asking the number of nighttime voids you had.
  Groups: Physical Activity and Sleep Study Controls
Other: Organ-Based — One in-person visit involving:
  Urethral vibratory sensation threshold Urethral Pressure Profilometry Cystometry Uroflowmetry Lidocaine Pre-Treatment Cystometry
  Groups: Organ-Based Study; Organ-Based Study Controls
Other: Qualitative Assessment of Patients with Urinary Urgency — Participation will include two interviews with a research assistant over the phone and are expected to take up to 60 minutes for each interview. The first interview will be done within four weeks from enrollment, before the start of treatment. The interview will include questions about participant's urinary urgency, including symptoms experienced, the onset of symptoms and other factors that affect urgency.
  Approximately three months after the start treatment the participant will be interviewed again. This interview will cover changes in symptoms and experience with treatment, such as side effects and satisfaction with treatment.
  Groups: Qualitative Assessment of Patients with Urinary Urgency Study

SUMMARY:
The purpose of this study is to define and characterize important subtypes of patients with urinary urgency to improve our understanding of the pathophysiology, risk factors, experiences, and comorbidities to lay the foundation for more effective treatment by focusing on the most bothersome and difficult to treat symptoms of urinary urgency and urgency urinary incontinence.

DETAILED DESCRIPTION:
LURN is pursuing deeper phenotyping of patients with urinary urgency and UUI using distinct, but related, projects. The Urinary Urgency Phenotyping Protocol is the overarching effort, and will comprise five integrated projects. Project A, the Observational Cohort, will be a large-scale accrual of male and female participants with urinary urgency and age-matched controls without any LUTS. Standardized clinical data, comprising information typically gathered at the patient clinic encounter, self-report symptom, urologic and non-urologic data, and biosamples will be collected. Using this group of participants, subsets will be identified for more focused and in-depth studies of urinary urgency and urgency incontinence. This more focused effort will be conducted as Project B: the Central Sensitization Study; Project C: the Physical Activity and Sleep Study; Project D: the Organ-Based Study; and Project E: the Qualitative Assessment of Patients with Urinary Urgency Study.

ELIGIBILITY:
Inclusion Criteria:

* Women or men presenting for evaluation or treatment of urinary urgency/ UUI to one of the LURN sites. These symptoms are not required to be the primary symptom(s) of presentation, but must be bothersome to the participant.
* Age ≥ 18 years.
* The presence of any of the urinary urgency or urgency incontinence symptoms based on responses to the LUTS Tool with a 1-month recall period (Appendix A) as follows:

Answered "sometimes", "often", or "always" on either:

* "During the past month, how often have you had a sudden need to rush to urinate?". Participants who answered "never" or "rarely" are not eligible since they are not deemed to have significant urinary urgency symptoms.
* "How often have you had a sudden need to rush to urinate for the fear of leaking urine?"
* Positive answer must also be associated with bother rating on that particular question of "somewhat", "quite a bit", or "a great deal"
* The ability to give informed consent and complete self-reported questionnaires electronically.
* Access to and willingness to utilize smart phone

Exclusion Criteria:

* a. Clinical impression of bladder outlet obstruction (based on symptoms or urodynamics) as primary etiology of LUTS.

  b. Gross hematuria/self-reported gross or visible urine in the blood. c. Significant neurologic disease or injury, including but not limited to: cerebral vascular accident with residual defect, Alzheimer's dementia, Parkinson's disease, traumatic brain injury, spinal cord injury, complicated spinal surgery, multiple sclerosis.

  d. Primary complaint is pelvic pain. e. Diagnosis of interstitial cystitis, chronic prostatitis, or chronic orchalgia.

  f. Pelvic or endoscopic GU surgery within the preceding 6 months (not including diagnostic cystoscopy).

  g. Ongoing symptomatic urethral stricture. h. History of LUT or pelvic malignancy. i. Current chemotherapy or other cancer therapy. j. Pelvic device or implant complication (e.g., sling or mesh complications). k. In men, prostate biopsy in the previous 6 months. l. In women, current pregnancy or planned pregnancy during the follow-up period.

  m. History of cystitis caused by tuberculosis, radiation therapy, or Cytoxan/cyclophosphamide therapy.

  n. Augmentation cystoplasty or cystectomy. o. Presence of urinary tract fistula. p. Current major psychiatric disorder or other psychiatric or medical issues that would interfere with study participation (e.g., dementia, psychosis, etc.).

  q. Inability to relay valid information, actively participate in the study, or provide informed consent (includes uncontrolled psychiatric disease).

  r. Difficulty reading or communicating in English. s. No access to internet/smart phone. t. Indwelling Foley catheter/routine self-catheterization. u. In addition to the criteria listed above, pregnancy during the study will be a study end point.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women with urinary urgency an/or urgency incontinence who are treatment-naïve patients, patients undergoing current treatment, and those who have failed therapies for lower urinary tract symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 840 (Estimated)
Dates: Start 2021-02-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in lower urinary tract symptoms | Baseline, 3 months, 6 month, 9 months,12 months
  Participants will be classified as treatment responders if they achieve at least a 10-point reduction from baseline on the OAB-q and/or respond "much better" or "very much better" on the PGI-I

SECONDARY OUTCOMES:
Examine the presence of sensory hypersensitivity in urinary urgency (with or without urgency incontinence) | Baseline
  Participants will rate pain intensity and unpleasantness on 0-100 numeric rating scales when ascending pressure is applied to the suprapubic area using a hand-held algometer
Assess the relationship between physical activity and sleep quality in men and women with bothersome urinary urgency | Baseline and 3 months
  Participants will wear a mobile tracker for two weeks at baseline and at 3 months to capture the average number of steps per 24 hours and number of nocturnal voids
The role of the urethra and its interaction with the bladder in LUT function and dysfunction | Baseline
  Urodynamic studies will be performed on urethra and bladder to assess urethral closure pressure, urethral sensation, and bladder volume

CONTACTS AND LOCATIONS:
Overall Officials: Henry Lai, MD, Study Chair — Washington University School of Medicine; John Graff, PhD, MS, Principal Investigator — Arbor Research Collaborative for Health - DCC
Locations (6):
- United States (6):
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Michigan, Ann Arbor, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Duke University, Durham, North Carolina
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
We do not plan to make IPD available.

REFERENCES:
- [Background] Cameron AP, Lewicky-Gaupp C, Smith AR, Helfand BT, Gore JL, Clemens JQ, Yang CC, Siddiqui NY, Lai HH, Griffith JW, Andreev VP, Liu G, Weinfurt K, Amundsen CL, Bradley CS, Kusek JW, Kirkali Z; Symptoms of Lower Urinary Tract Dysfunction Research Network Study Group. Baseline Lower Urinary Tract Symptoms in Patients Enrolled in LURN: A Prospective, Observational Cohort Study. J Urol. 2018 Apr;199(4):1023-1031. doi: 10.1016/j.juro.2017.10.035. Epub 2017 Oct 28. PMID 29111381
- [Background] Weinfurt KP, Griffith JW, Flynn KE, Cella D, Bavendam T, Wiseman JB, Andreev VP, Lai HH, Liu AB, Kirkali Z, Cameron AP, Bradley CS; LURN Study Group. The Comprehensive Assessment of Self-Reported Urinary Symptoms: A New Tool for Research on Subtypes of Patients with Lower Urinary Tract Symptoms. J Urol. 2019 Jun;201(6):1177-1183. doi: 10.1097/JU.0000000000000140. PMID 30730410
- [Background] Andreev VP, Liu G, Yang CC, Smith AR, Helmuth ME, Wiseman JB, Merion RM, Weinfurt KP, Cameron AP, Lai HH, Cella D, Gillespie BW, Helfand BT, Griffith JW, DeLancey JOL, Fraser MO, Clemens JQ, Kirkali Z; LURN Study Group. Symptom Based Clustering of Women in the LURN Observational Cohort Study. J Urol. 2018 Dec;200(6):1323-1331. doi: 10.1016/j.juro.2018.06.068. Epub 2018 Jul 7. PMID 29990467
- [Background] Reynolds WS, Dmochowski R, Wein A, Bruehl S. Does central sensitization help explain idiopathic overactive bladder? Nat Rev Urol. 2016 Aug;13(8):481-91. doi: 10.1038/nrurol.2016.95. Epub 2016 Jun 1. PMID 27245505
- [Background] Ge TJ, Vetter J, Lai HH. Sleep Disturbance and Fatigue Are Associated With More Severe Urinary Incontinence and Overactive Bladder Symptoms. Urology. 2017 Nov;109:67-73. doi: 10.1016/j.urology.2017.07.039. Epub 2017 Aug 4. PMID 28826875
- [Derived] Hokanson JA, DeLancey JOL, Kirby AC, Gillespie B, Lai HH, Kreder KJ, Bretschneider CE, Slavik N, Andrews C, Andreev V, Black L, Richardson S, Kenton K, Kirkali Z, Yang CC; Symptoms of Lower Urinary Tract Dysfunction Research Network (LURN) Study Group. Expanded Physiological Testing of the Lower Urinary Tract in Asymptomatic Women and Those With Urgency Urinary Incontinence: Findings From the LURN-Organ Study. Neurourol Urodyn. 2025 Jun;44(5):987-996. doi: 10.1002/nau.70038. Epub 2025 Mar 31. PMID 40159923
- See also: Study website — http://nih-lurn.org